CLINICAL TRIAL: NCT00003445
Title: Neoadjuvant Chemotherapy With Docetaxel in Advanced Cervical Carcinoma
Brief Title: Docetaxel in Treating Patients With Advanced Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Oncologico Cooperativo del Sur (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: GOCS-04-CC-97; CDR0000066473 (Registry Identifier: PDQ (Physician Data Query)); NCI-V98-1456
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2001-09

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IIB cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of docetaxel in treating patients with advanced cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the antitumor activity of docetaxel as neoadjuvant chemotherapy in patients with locally advanced squamous cell carcinoma of the cervix. II. Assess the tumor response, toxic effect, and survival rate of this regimen in these patients.

OUTLINE: Patients receive docetaxel IV over 1 hour on day 1. Treatment is repeated every 3 weeks for 3 courses. Patients are followed every 3 months posttreatment.

PROJECTED ACCRUAL: A total of 16-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IIB, IIIA, IIIB, and IVA squamous cell carcinoma of the cervix Bidimensionally measurable disease No bilateral hydronefrosis

PATIENT CHARACTERISTICS: Age: Any age Performance status: WHO 0-2 Life expectancy: At least 12 weeks Hematopoietic: Hemoglobin at least 10 g/dL Leukocytes at least 4,000/mm3 Platelet count at least 75,000/mm3 Hepatic: Bilirubin less than 1.25 times upper limit of normal (ULN) AST less than 1.25 times ULN Renal: BUN less than 30 mg/dL AND Creatinine less than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: No prior or other concurrent malignancies, other than properly treated basal cell skin cancer

PRIOR CONCURRENT THERAPY: Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-12; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Teodoro Vallejo, MD, Study Chair — Grupo Oncologico Cooperativo del Sur
Locations (1):
- Unidad Oncologica Del Comahue, Neuquén, Argentina